CLINICAL TRIAL: NCT02752620
Title: Osteopathic Manipulative Treatment Versus Therapeutic Exercises in Subjects With Chronic Non-specific Low Back Pain: a Randomized Controlled and Double-blind Trial
Brief Title: Osteopathic Manipulative Treatment Versus Therapeutic Exercises in Subjects With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Estácio S.A. (Other)
Responsible Party: Principal Investigator, Frederico de Oliveira Meirelles, MEIRELLES, F. O., Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 46194215.9.0000.5284
Record Dates: First submitted 2016-04-23; First posted 2016-04-27 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Low Back Pain
Keywords: osteopathic manipulative treatment; Chronic nonspecific low back pain; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): We selected two types of osteopathic techniques for this study:
  Technical articulation: rhythmic technique with low speed in which the goal is the full gain range of motion.
  Myofascial techniques (Neuromuscular): techniques involving lateral stretching, linear, deep pressures and pulls of the origins and insertions aiming at a myofascial relaxation.
  Sacroiliac articulatory technique; Dorsal articulatory technique; Lumbar paraspinal muscles stretching technique; Lumbar myofascial technique (inhibitory).
  Interventions: Other: Osteopathic Manipulative Treatment
- Exercise Therapy (Active Comparator): 2 types of therapeutic exercises techniques were used:
  * Stabilization exercises
  * Stretches
  Stabilization exercises:
  Bridge on the ball 10 - 15 sec Side plank 10 - 15 sec Front board 10 - 15 sec active mobilization lumbopelvic 3 x 6 rep Squats with the ball on the wall 3 x 8 rep
  Static-passive stretch (2 x 30 sec):
  Paraspinal; Abdominals; Quadratus lumborum; Hip extenders; Hip flexors; Hip abductors; Hip adductors.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment
  Arms: Osteopathic Manipulative Treatment
Other: Exercise Therapy
  Arms: Exercise Therapy

SUMMARY:
This study evaluates the effectiveness of treatment osteopathic manipulation in the treatment of subjects with chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with constant or intermittent low back pain with intensity greater than 30 mm visual analog scale (VAS) for at least three months duration, with a diagnosis of chronic low back pain

Exclusion Criteria:

* Subjects who have spine fractures,
* Dislocations
* Ligament ruptures
* Muscle ruptures
* Skin lacerations
* Sacroiliitis
* Vertebral osteomyelitis
* Infection
* Disc herniations with radicular symptoms
* Rheumatic disorders
* Cauda equina syndrome
* Tumors
* Referred pain visceral
* Red flags
* Lower limb discrepancy greater than 2 cm
* Several conditions requiring participants to be absent for more than two weeks of activities in the experiment
* Positioning itself as not volunteer the same.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pain | 5 weeks
  VAS (VISUAL ANALOGUE SCALE)

SECONDARY OUTCOMES:
Disability | 5 weeks
  Oswestry Disability Index 2.0
kinesiophobia | 5 weeks
  Tampa Scale for Kinesiophobia
Depression | 5 weeks
  Beck Scale for Depression

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Meirelles, Master /PT, Principal Investigator — UERJ
Locations (1):
- Estácio de Sá University, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No